CLINICAL TRIAL: NCT02458313
Title: Nicotinic Agonist Effects on BMI and Neuronal Response in Overweight/Obese Adults
Brief Title: Nicotinic Agonist Effects on BMI and Neuronal Response
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 15-0650; UL1TR001082 (NIH)
Record Dates: First submitted 2015-05-21; First posted 2015-06-01 (Estimated); Results first posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — 3-(2,4-dimethoxybenzylidene)anabaseine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DMXB-A (Experimental): 150 mg DMXB-A (3-(2,4-dimethoxybenzylidene anabaseine) b.i.d. for 12 weeks.
  Interventions: Drug: DMXB-A
- Placebo (Placebo Comparator): Placebo capsules b.i.d. for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: DMXB-A — 150 mg DMXB-A (3-(2,4-dimethoxybenzylidene anabaseine) b.i.d. for 12 weeks.
  Other Names: 3-(2,4-dimethoxybenzylidene anabaseine
  Arms: DMXB-A
Other: Placebo — Placebo capsules b.i.d. for 12 weeks
  Arms: Placebo

SUMMARY:
Obesity is a serious and growing health problem in the United States. Obesity is associated with health problems such as type-2 diabetes and cardiovascular disease, leading to decreased quality of life and increased mortality. Given the health and quality-of-life effects of obesity, developing effective treatments clearly is an important goal.

This study plans to learn more about the effects of an investigational new drug (DMXB-A (3-(2,4-dimethoxybenzylidene anabaseine)) and its effects on obesity. The study drug has similar effects to nicotine. Since nicotine has been found to affect appetite, the investigators are interested in studying effects of the study drug, which has some similarities to nicotine, on how your brain responds to such things as pictures of food. The study drug has not been approved by the Food and Drug Administration (FDA), and is considered experimental.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/obese (BMI > 27)
* Between 21-65 years old

Exclusion Criteria:

* Known cardiovascular disease (e.g., coronary artery disease, uncontrolled hypertension
* Women capable of conception (must be post-menopausal, surgically sterilized, or have adhered to an anti-contraception birth control regimen for at least 1 year)
* Nicotine use
* Significant endocrine/metabolic disease
* Kidney disease
* Neurological illness
* Liver disease
* Medication use affecting appetite and/or metabolism
* MRI-specific exclusion criteria (e.g., claustrophobia, metal in the body)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Tregellas, Ph.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via flyer and email advertisement in Aurora, CO, between April 2016 and November 2021.
Period: Overall Study
Arm/Group | DMXB-A | Placebo
Started | 30 | 31
Completed | 23 | 21
Not Completed | 7 | 10
Not completed — Withdrawal by Subject | 6 | 8
Not completed — Excluded for motion during MRI | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DMXB-A | Placebo | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.17 (11.27) | 43.71 (11.06) | 43.93 (11.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 45
  Male | 7 | 9 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 7 | 9
  Not Hispanic or Latino | 28 | 24 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 2 | 9
  White | 22 | 26 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 31 | 61

OUTCOME MEASURES:

1. Primary Outcome: Neuronal Response to Visual Food Cues
Description: Neuronal response (insula) while viewing visual food cues
Time Frame: 14 weeks
Measure: Mean (Standard Deviation); unit: % BOLD signal
Arm/Group | DMXB-A | Placebo
Number analyzed (Participants) | 23 | 21
% BOLD signal
  Baseline | .035 (.073) | .045 (.095)
  Post-intervention | .029 (.094) | .019 (.094)
Statistical Analysis 1: Comparison: DMXB-A vs Placebo; Test type: Superiority — DMXB-A vs. Placebo groups compared at baseline; p = 0.647, t-test, 2 sided
Statistical Analysis 2: Comparison: DMXB-A vs Placebo; DMXB-A vs. Placebo groups compared post-intervention; Test type: Superiority; p = 0.679, t-test, 2 sided

2. Primary Outcome: Resting-state Neuronal Response
Description: Neuronal response (default mode network) during rest
Time Frame: 14 weeks
Measure: Mean (Standard Deviation); unit: Percent BOLD signal
Arm/Group | DMXB-A | Placebo
Number analyzed (Participants) | 23 | 21
Percent BOLD signal
  Baseline | 2.008 (.072) | 2.009 (.064)
  Post-intervention | 1.991 (.106) | 1.995 (.076)
Statistical Analysis 1: Comparison: DMXB-A vs Placebo; DMXB-A vs. Placebo groups compared at baseline; Test type: Superiority; p = 0.951, t-test, 2 sided
Statistical Analysis 2: Comparison: DMXB-A vs Placebo; DMXB-A vs. Placebo groups compared post-intervention; Test type: Superiority; p = 0.884, t-test, 2 sided

3. Secondary Outcome: Body Weight
Description: Body weight
Time Frame: 14 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Fat Mass
Description: Fat mass
Time Frame: 14 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Appetite Rating
Description: Hunger ratings via VAS scale (0-100)
Time Frame: 14 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data collected at weeks 2, 4, 6, 8, and 10 of the intervention, and at the post-intervention visit, up to 14 weeks.
Arm/Group | DMXB-A | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 16/30 | 18/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DMXB-A (N=30) | Placebo (N=31)
Fever (General disorders) | 2 (2) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 3 (7) | 4 (5)
Body aches (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Dry mouth (General disorders) | 1 (1) | 4 (6)
Increased thirst (General disorders) | 0 (0) | 2 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acid reflux (Gastrointestinal disorders) | 0 (0) | 1 (1)
Insomnia (General disorders) | 1 (1) | 3 (4)
Bad breath (General disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sore throat (General disorders) | 3 (3) | 1 (1)
Congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Drowsiness (General disorders) | 1 (2) | 1 (1)
Change in appetite (Metabolism and nutrition disorders) | 1 (1) | 5 (7)
Nausea (Gastrointestinal disorders) | 7 (9) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 4 (6) | 4 (6)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pink eye (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 1 (1)
Abdominal pain (General disorders) | 1 (1) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 1 (1)
Forgetful (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/13/NCT02458313/Prot_SAP_000.pdf